CLINICAL TRIAL: NCT05975840
Title: A Phase I/II Observer-blind, Randomized, Multi-center Trial to Evaluate the Safety and Immunogenicity of Different Formulations of Monovalent Influenza A/Astrakhan/3212/2020 Like (H5N8) Virus Vaccine With AS03 Adjuvant System (Referred to as Q-Pan H5N8), Given as a Two-dose Series to Adults 18 to 64 Years of Age and 65 Years of Age and Older
Brief Title: Safety and Immunogenicity of Different Formulations of Monovalent Influenza A/Astrakhan/3212/2020 Like (H5N8) Virus Vaccine With AS03 Adjuvant System in Medically Stable Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 219833
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Influenza, Human
Keywords: Influenza; Safety; Immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be observer blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Age group 18-64: FLU Q-PAN H5N8 375_B (Active Comparator): Participants received 2 doses of 375_B vaccine formulation, 21 days apart.
  Interventions: Biological: FLU Q-PAN H5N8 375_B
- Age group 18-64: FLU Q-PAN H5N8 375_A (Active Comparator): Participants received 2 doses of 375_A vaccine formulation, 21 days apart.
  Interventions: Biological: FLU Q-PAN H5N8 375_A
- Age group 18-64: FLU Q-PAN H5N8 750_B (Active Comparator): Participants received 2 doses of 750_B vaccine formulation, 21 days apart.
  Interventions: Biological: FLU Q-PAN H5N8 750_B
- Age group 18-64: FLU Q-PAN H5N8 750_A (Active Comparator): Participants received 2 doses of 750_A vaccine formulation, 21 days apart.
  Interventions: Biological: FLU Q-PAN H5N8 750_A
- Age group >=65: FLU Q-PAN H5N8 375_B (Active Comparator): Participants received 2 doses of 375_B vaccine formulation, 21 days apart.
  Interventions: Biological: FLU Q-PAN H5N8 375_B
- Age group >=65: FLU Q-PAN H5N8 375_A (Active Comparator): Participants received 2 doses of 375_A vaccine formulation, 21 days apart.
  Interventions: Biological: FLU Q-PAN H5N8 375_A
- Age group >=65: FLU Q-PAN H5N8 750_B (Active Comparator): Participants received 2 doses of 750_B vaccine formulation, 21 days apart.
  Interventions: Biological: FLU Q-PAN H5N8 750_B
- Age group >=65: FLU Q-PAN H5N8 750_A (Active Comparator): Participants received 2 doses of 750_A vaccine formulation, 21 days apart.
  Interventions: Biological: FLU Q-PAN H5N8 750_A

INTERVENTIONS:
Biological: FLU Q-PAN H5N8 375_B — Participants received 2 doses of 375_B vaccine formulation by intramuscular injection in the non-dominant arm.
  Arms: Age group 18-64: FLU Q-PAN H5N8 375_B; Age group >=65: FLU Q-PAN H5N8 375_B
Biological: FLU Q-PAN H5N8 375_A — Participants received 2 doses of 375_A vaccine formulation by intramuscular injection in the non-dominant arm.
  Arms: Age group 18-64: FLU Q-PAN H5N8 375_A; Age group >=65: FLU Q-PAN H5N8 375_A
Biological: FLU Q-PAN H5N8 750_B — Participants received 2 doses of 750_B vaccine formulation by intramuscular injection in the non-dominant arm.
  Arms: Age group 18-64: FLU Q-PAN H5N8 750_B; Age group >=65: FLU Q-PAN H5N8 750_B
Biological: FLU Q-PAN H5N8 750_A — Participants received 2 doses of 750_A vaccine formulation by intramuscular injection in the non-dominant arm.
  Arms: Age group 18-64: FLU Q-PAN H5N8 750_A; Age group >=65: FLU Q-PAN H5N8 750_A

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of different formulations of monovalent Influenza A/Astrakhan/3212/2020-like virus vaccine with AS03 adjuvant system in adults greater than or equal to (>=)18 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable participants as established by medical history and clinical examination before entering into the study.
* A male or female >=18 years of age at the time of signing consent form.
* Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participant prior to performance of any study specific procedure.
* Female participants of childbearing potential or non-childbearing potential may be enrolled in the study if specific criteria are met.

Exclusion Criteria:

* Current diagnosis or history of autoimmune disorder(s) except hypothyroidism due to Hashimoto's thyroiditis.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Clinically significant acute or chronic pulmonary, cardiovascular, hepatic, or renal disease that appears uncontrolled or untreated, as determined by history or physical examination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history, physical examination, or abnormalities in screening blood tests.
* Recurrent history of or uncontrolled neurological disorders or seizures.
* History of Guillain-Barré syndrome.
* Diagnosed with cancer, or treatment for cancer within 3 years.

  * Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
  * Persons with a history of histologically confirmed basal cell carcinoma of the skin successfully treated with local excision only, are accepted and are eligible, but other histologic types of skin cancer are exclusionary.
  * Women who are disease-free 3 years or more after treatment for breast cancer and receiving long-term prophylaxis are eligible.
* Documented human immunodeficiency virus-positive participants.
* Bedridden participants.
* Personal or family history of narcolepsy.
* Food and Drug Administration (FDA) toxicity Grade 2, or greater, laboratory tests at Screening.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* Use of any investigational or non-registered product other than the study vaccine during the period beginning 30 days before the first dose of study vaccine (Day -29 to Day 1), or planned use during the entire study period.
* Use of public health emergency vaccines like coronavirus disease 2019 (COVID-19), Monkey pox (mpox) etc. These can be given at any time, but there should a gap of 2 - weeks before a dose of study vaccine can be given.
* Use of any licensed vaccines: prior to receipt of the study vaccine and continuing up to 3 weeks after receiving the dose 2 of study vaccine.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the first dose of study vaccine or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first vaccine dose and through the entire study period. For corticosteroids, this will mean prednisone equivalent >=20 milligrams/day for 14 days or a total of >=280 mg of prednisone equivalent dose in any 14-day period. Inhaled and topical steroids are allowed.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within 2 months after completion of the vaccination series.
* History of/or current drug/alcohol abuse.
* Any study personnel or their immediate dependents, family, or household member.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non investigational vaccine/product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Chamblee, Georgia
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, El Dorado, Kansas
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Started | 66 | 65 | 64 | 63 | 66 | 64 | 66 | 64
Completed | 61 | 52 | 59 | 59 | 61 | 61 | 62 | 58
Not Completed | 5 | 13 | 5 | 4 | 5 | 3 | 4 | 6
Not completed — Other | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 6 | 3 | 1 | 4 | 1 | 2 | 4
Not completed — Migrated/moved from the study area | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 2 | 2 | 0 | 2 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population comprised of Exposed analysis set who received at least 1 dose of study vaccine. Summary of "Race/Ethnicity, Customized" baseline categorical variables are presented as de-identified to prevent risk of participant re-identification.
Groups:
- Total: Total of all reporting groups
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A | Total
Number analyzed (Participants) | 66 | 65 | 64 | 63 | 66 | 64 | 66 | 64 | 518
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Based on Food and Drug Administration (FDA) immunogenicity criteria for influenza vaccines, age continuous is presented based on the age categories of 18-64 and 65 and above years of age.
  Years
    18-64 Years of age: number analyzed (Participants) | 66 | 65 | 64 | 63 | 0 | 0 | 0 | 0 | 258
    18-64 Years of age | 42.5 (13.5) | 42.3 (12.3) | 40.7 (12.8) | 44.0 (13.4) |  |  |  |  | 42.4 (13.0)
    >=65 Years of age: number analyzed (Participants) | 0 | 0 | 0 | 0 | 66 | 64 | 66 | 64 | 260
    >=65 Years of age |  |  |  |  | 70.9 (4.7) | 71.9 (5.4) | 72.1 (5.2) | 71.0 (5.2) | 71.5 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 24 | 29 | 40 | 35 | 32 | 41 | 36 | 271
  Male | 32 | 41 | 35 | 23 | 31 | 32 | 25 | 28 | 247
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 41 | 39 | 38 | 54 | 50 | 52 | 47 | 355
  Other, combined to maintain patient confidentiality | 32 | 24 | 25 | 25 | 12 | 14 | 14 | 17 | 163

OUTCOME MEASURES:

1. Primary Outcome: Hemagglutination-inhibiting (HI) Antibody Titers Against Vaccine-homologous H5N8
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: At Day 43
Population: Analysis was performed on the Per-protocol set (PPS) which included all eligible participants who received the 2 doses of study intervention as per protocol, had Day 1 and Day 43 post dose anti-HI immunogenicity results as per blood draw interval at Day 43. Only those participants with data available at the specified timepoint have been analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 56 | 46 | 47 | 49 | 47 | 40 | 43 | 44
Titer | 117.5 [97.0 to 141.8] | 175.2 [142.2 to 216.0] | 121.8 [99.2 to 150.1] | 176.6 [144.2 to 216.2] | 80.6 [64.3 to 101.1] | 110.2 [85.3 to 139.7] | 84.0 [66.6 to 107.0] | 129.3 [102.7 to 164.1]

2. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Serum HI Antibody Titers Against Vaccine-homologous H5N8
Description: The GMFR is defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus.
Time Frame: At Day 43
Population: PPS population. Only those participants with data available at the specified timepoint have been analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 56 | 46 | 47 | 49 | 47 | 40 | 43 | 44
Ratio | 21.7 [18.3 to 26.7] | 33.0 [26.8 to 40.7] | 23.7 [18.7 to 28.3] | 33.1 [27.2 to 40.7] | 11.7 [9.3 to 14.6] | 14.3 [12.3 to 20.2] | 12.8 [9.6 to 15.4] | 19.5 [14.8 to 23.7]

3. Primary Outcome: Number of Seroprotected (SP) Participants for HI Antibody Titers
Description: Seroprotection rate is defined as the number of participants with HI titer value greater than or equal to (>=) 1:40 which is considered as indicating protection.
Time Frame: At Day 43
Population: PPS population. Only those participants with data available at the specified timepoint have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 56 | 46 | 47 | 49 | 47 | 40 | 43 | 44
Participants | 56 | 45 | 46 | 49 | 43 | 37 | 41 | 41

4. Primary Outcome: Number of Participants Reporting Each Solicited Administration Site Event Following Dose 1
Description: Solicited administration site events included pain, redness and swelling.
Time Frame: 7 days (Day 1 to Day 7) following dose 1
Population: The analysis was performed on the Diary Set for dose 1 (DS1) which included participants who received a study intervention and provided information on at least 1 solicited adverse event (AE) on at least 1 day.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 65 | 59 | 62 | 63 | 64 | 63 | 64 | 64
Participants
  Pain | 39 | 34 | 27 | 38 | 23 | 22 | 14 | 29
  Redness | 3 | 0 | 2 | 2 | 0 | 1 | 0 | 4
  Swelling | 2 | 0 | 2 | 2 | 2 | 1 | 0 | 5

5. Primary Outcome: Number of Participants Reporting Each Solicited Administration Site Event Following Dose 2
Description: Solicited administration site events included pain, redness and swelling.
Time Frame: 7 days (Day 22 to Day 28) following dose 2
Population: Analysis was performed on the DS2 which included participants who received a study intervention and provided information on at least 1 solicited AE on at least 1 day.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 63 | 52 | 53 | 55 | 49 | 45 | 49 | 49
Participants
  Pain | 31 | 19 | 21 | 24 | 17 | 14 | 12 | 15
  Redness | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 3
  Swelling | 3 | 0 | 1 | 1 | 0 | 1 | 0 | 2

6. Primary Outcome: Number of Participants Reporting Each Solicited Systemic Event Following Dose 1
Description: Solicited systemic events included fatigue, fever, headache, muscle ache, joint pain, shivering (chills), sweating, gastrointestinal symptoms (nausea, vomiting, diarrhea, abdominal pain). Fever is defined as temperature >=38 degrees Celsius (°C) for oral route (preferred location for measuring temperature).
Time Frame: 7 days (Day 1 to Day 7) following dose 1
Population: DS1 population
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 65 | 59 | 62 | 63 | 64 | 63 | 64 | 64
Participants
  Fatigue | 25 | 18 | 15 | 20 | 9 | 13 | 6 | 12
  Fever | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Headache | 19 | 12 | 10 | 15 | 9 | 12 | 5 | 12
  Muscle ache | 23 | 22 | 15 | 26 | 9 | 12 | 8 | 16
  Joint pain | 12 | 9 | 3 | 9 | 2 | 9 | 4 | 6
  Shivering (chills) | 6 | 7 | 1 | 5 | 5 | 2 | 0 | 4
  Sweating | 10 | 7 | 3 | 7 | 6 | 2 | 2 | 4
  Nausea | 11 | 6 | 4 | 7 | 5 | 2 | 5 | 4
  Vomiting | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Diarrhea | 7 | 4 | 6 | 5 | 2 | 1 | 4 | 3
  Abdominal pain | 6 | 3 | 2 | 4 | 7 | 3 | 5 | 4

7. Primary Outcome: Number of Participants Reporting Each Solicited Systemic Event Following Dose 2
Description: as for outcome 6
Time Frame: 7 days (Day 22 to Day 28) following dose 2
Population: DS2 population
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 63 | 52 | 53 | 55 | 49 | 45 | 49 | 49
Participants
  Fatigue | 18 | 9 | 10 | 11 | 5 | 12 | 4 | 8
  Fever | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1
  Headache | 19 | 6 | 4 | 10 | 5 | 4 | 4 | 5
  Muscle ache | 17 | 10 | 10 | 15 | 6 | 7 | 3 | 7
  Joint pain | 8 | 6 | 3 | 6 | 3 | 1 | 2 | 4
  Shivering (chills) | 3 | 2 | 3 | 3 | 1 | 1 | 1 | 1
  Sweating | 5 | 3 | 3 | 5 | 4 | 2 | 0 | 1
  Nausea | 2 | 2 | 0 | 6 | 1 | 3 | 1 | 2
  Vomiting | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0
  Diarrhea | 6 | 3 | 3 | 3 | 1 | 1 | 2 | 1
  Abdominal pain | 2 | 2 | 2 | 6 | 1 | 1 | 1 | 1

8. Primary Outcome: Number of Participants With Any Increase in Toxicity Grading in Hematological Laboratory Parameters Following Dose 1
Description: Hemoglobin, white blood cells (WBC) increase, WBC decrease, platelets, neutrophils, lymphocytes and eosinophils were graded by FDA toxicity grading scale in which grades are Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe and Grade 4 = potentially life threatening. Blood samples were collected for safety laboratory tests from the first 50% of participants of each age and dose group, at 7 days following each vaccination (i.e., Visit 2 and Visit 4).
Time Frame: 7 days (Day 1 to Day 7) following dose 1
Population: Analysis was performed on the Exposed set for dose 1 (ES1), which included participants who received a study intervention and for whom blood samples were collected and analyzed for the safety laboratory tests, at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 33 | 34 | 33 | 32 | 32 | 36 | 35 | 36
Participants
  Hemoglobin | 2 | 5 | 1 | 6 | 7 | 6 | 7 | 7
  WBC Increase: number analyzed (Participants) | 33 | 34 | 33 | 32 | 32 | 36 | 34 | 35
  WBC Increase | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1
  WBC Decrease: number analyzed (Participants) | 33 | 34 | 33 | 32 | 32 | 36 | 34 | 35
  WBC Decrease | 2 | 2 | 0 | 3 | 0 | 1 | 1 | 0
  Platelets: number analyzed (Participants) | 33 | 33 | 33 | 32 | 32 | 35 | 35 | 36
  Platelets | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Neutrophils Absolute | 3 | 1 | 2 | 3 | 0 | 2 | 1 | 1
  Lymphocytes Absolute | 0 | 1 | 0 | 0 | 0 | 5 | 1 | 0
  Eosinophils Absolute: number analyzed (Participants) | 31 | 33 | 32 | 30 | 32 | 35 | 33 | 36
  Eosinophils Absolute | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

9. Primary Outcome: Number of Participants With Any Increase in Toxicity Grading in Hematological Laboratory Parameters Following Dose 2
Description: Hemoglobin, WBC increase, WBC decrease, platelets, neutrophils, lymphocytes and eosinophils were graded by FDA toxicity grading scale in which grades are Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe and Grade 4 = potentially life threatening. Blood samples were collected for safety laboratory tests from the first 50% of participants of each age and dose group, at 7 days following each vaccination (i.e., Visit 2 and Visit 4).
Time Frame: 7 days (Day 22 to Day 28) following dose 2
Population: Analysis was performed on the Exposed set for dose 2 (ES2), which included participants who received a study intervention and for whom blood samples were collected and analyzed for the safety laboratory tests, at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 31 | 24 | 29 | 28 | 23 | 23 | 22 | 23
Participants
  Hemoglobin | 5 | 3 | 3 | 2 | 2 | 4 | 3 | 4
  WBC Increase: number analyzed (Participants) | 31 | 24 | 28 | 27 | 23 | 23 | 21 | 22
  WBC Increase | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 2
  WBC Decrease: number analyzed (Participants) | 31 | 24 | 28 | 27 | 23 | 23 | 21 | 22
  WBC Decrease | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Platelets | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophils Absolute: number analyzed (Participants) | 31 | 24 | 29 | 28 | 23 | 23 | 22 | 22
  Neutrophils Absolute | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  Lymphocytes Absolute: number analyzed (Participants) | 31 | 24 | 29 | 28 | 23 | 23 | 22 | 22
  Lymphocytes Absolute | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1
  Eosinophils Absolute: number analyzed (Participants) | 30 | 24 | 26 | 25 | 22 | 22 | 21 | 22
  Eosinophils Absolute | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0

10. Primary Outcome: Number of Participants With Any Increase in Toxicity Grading in Biochemical Laboratory Parameters Following Dose 1
Description: Sodium increase, sodium decrease, potassium increase, potassium decrease, creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, total bilirubin and blood urea nitrogen (BUN) were graded by FDA toxicity grading scale in which grades are Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe and Grade 4 = potentially life threatening. Blood samples were collected for safety laboratory tests from the first 50% of participants of each age and dose group, at 7 days following each vaccination (i.e., Visit 2 and Visit 4).
Time Frame: 7 days (Day 1 to Day 7) following dose 1
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 33 | 34 | 33 | 33 | 34 | 36 | 35 | 36
Participants
  Sodium Increase | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0
  Sodium Decrease | 2 | 3 | 3 | 1 | 4 | 4 | 5 | 4
  Potassium Increase | 1 | 1 | 6 | 1 | 5 | 7 | 2 | 5
  Potassium Decrease | 1 | 1 | 4 | 1 | 0 | 0 | 1 | 4
  Creatinine | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  ALT: number analyzed (Participants) | 33 | 34 | 33 | 32 | 33 | 36 | 35 | 36
  ALT | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 2
  AST | 0 | 1 | 2 | 0 | 0 | 0 | 3 | 4
  Alkaline Phosphatase | 1 | 3 | 2 | 0 | 4 | 3 | 2 | 3
  Total Bilirubin: number analyzed (Participants) | 29 | 30 | 32 | 29 | 33 | 35 | 34 | 36
  Total Bilirubin | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  BUN | 0 | 1 | 0 | 0 | 2 | 5 | 4 | 2

11. Primary Outcome: Number of Participants With Any Increase in Toxicity Grading in Biochemical Laboratory Parameters Following Dose 2
Description: Sodium increase, sodium decrease, potassium increase, potassium decrease, creatinine, ALT, AST, alkaline phosphatase, total bilirubin and BUN were graded by FDA toxicity grading scale in which grades are Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe and Grade 4 = potentially life threatening. Blood samples were collected for safety laboratory tests from the first 50% of participants of each age and dose group, at 7 days following each vaccination (i.e., Visit 2 and Visit 4).
Time Frame: 7 days (Day 22 to Day 28) following dose 2
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 32 | 26 | 29 | 28 | 24 | 23 | 22 | 23
Participants
  Sodium Increase | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Sodium Decrease | 1 | 2 | 1 | 2 | 1 | 2 | 2 | 1
  Potassium Increase | 2 | 1 | 1 | 1 | 4 | 1 | 4 | 3
  Potassium Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Creatinine | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  ALT: number analyzed (Participants) | 32 | 26 | 29 | 27 | 23 | 23 | 22 | 23
  ALT | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0
  AST: number analyzed (Participants) | 30 | 26 | 29 | 28 | 24 | 23 | 22 | 23
  AST | 1 | 0 | 1 | 1 | 0 | 1 | 4 | 0
  Alkaline Phosphatase | 1 | 3 | 0 | 0 | 3 | 2 | 2 | 3
  Total Bilirubin: number analyzed (Participants) | 31 | 26 | 26 | 25 | 24 | 23 | 21 | 22
  Total Bilirubin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BUN | 1 | 1 | 0 | 0 | 1 | 3 | 1 | 5

12. Primary Outcome: Number of Participants Reporting Unsolicited AEs Following Dose 1
Description: An unsolicited adverse event is defined as an adverse event that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Time Frame: 21 days (Day 1 to Day 22) following dose 1
Population: Analysis was performed on the total ES population that reported unsolicited AEs for dose 1 at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 66 | 65 | 64 | 63 | 66 | 64 | 66 | 64
Participants | 4 | 6 | 7 | 7 | 4 | 5 | 5 | 8

13. Primary Outcome: Number of Participants Reporting Unsolicited AEs Following Dose 2
Description: as for outcome 12
Time Frame: 21 days (Day 22 to Day 43) following dose 2
Population: Analysis was performed on the total ES population that reported unsolicited AEs for dose 2 at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 63 | 52 | 54 | 55 | 49 | 45 | 49 | 49
Participants | 3 | 4 | 2 | 3 | 6 | 3 | 3 | 1

14. Primary Outcome: Number of Participants Reporting Unsolicited Medically Attended Adverse Events (MAEs) Following Dose 1
Description: MAE is defined as an AE that results in an unscheduled visit to a medical professional (e.g., symptoms or illnesses requiring a hospitalization, emergency room visit, or visit to/by a healthcare provider).
Time Frame: 21 days (Day 1 to Day 22) following dose 1
Population: Analysis was performed on the total ES population that reported unsolicited MAEs for dose 1 at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 66 | 65 | 64 | 63 | 66 | 64 | 66 | 64
Participants | 1 | 3 | 3 | 3 | 2 | 1 | 1 | 3

15. Primary Outcome: Number of Participants Reporting Unsolicited MAEs Following Dose 2
Time Frame: 21 days (Day 22 to Day 43) following dose 2
Population: Analysis was performed on the total ES population that reported unsolicited MAEs for dose 2 at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 63 | 52 | 54 | 55 | 49 | 45 | 49 | 49
Participants | 2 | 1 | 1 | 2 | 1 | 0 | 2 | 0

16. Primary Outcome: Number of Participants Reporting Unsolicited MAEs up to 6 Months Post Dose 2 (Administered on Day 22)
Time Frame: Up to 6 months post dose 2 (administered on Day 22)
Population: Analysis was performed on the total ES population that reported unsolicited MAEs for dose 2 at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 66 | 65 | 64 | 63 | 66 | 64 | 66 | 64
Participants | 4 | 6 | 6 | 8 | 6 | 6 | 11 | 8

17. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) up to Day 43
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an abnormal pregnancy outcome (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy), or is a suspected transmission of any infectious agent via an authorized medicinal product.
Time Frame: From Day 1 to Day 43
Population: The analysis was performed on the Total ES which included participants who received a study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 66 | 65 | 64 | 63 | 66 | 64 | 66 | 64
Participants | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 1

18. Primary Outcome: Number of Participants Reporting SAEs up to 6 Months Post Dose 2 (Administered on Day 22)
Time Frame: Day 1 to 6 months post dose 2 (administered on Day 22)
Population: The analysis was performed on the Total ES which included participants who received a study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 66 | 65 | 64 | 63 | 66 | 64 | 66 | 64
Participants | 1 | 1 | 0 | 2 | 2 | 2 | 2 | 2

19. Primary Outcome: Number of Participants Reporting Potential Immune-mediated Diseases (pIMDs) up to Day 43
Description: pIMDs are defined a subset of AEs of special interest that includes autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: From Day 1 to Day 43
Population: The analysis was performed on the Total ES which included participants who received a study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 66 | 65 | 64 | 63 | 66 | 64 | 66 | 64
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: HI Antibody Titers Against Vaccine-homologous H5N8
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Day 1, Day 22, and 6 months post dose 2 (administered on Day 22)
Population: PPS population. Only those participants with data available at the specified time points have been analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 64 | 62 | 59 | 56 | 62 | 56 | 60 | 60
Titer
  Day 1 | 5.4 [5.0 to 5.8] | 5.2 [5.0 to 5.5] | 5.2 [5.0 to 5.4] | 5.4 [4.9 to 5.9] | 6.7 [5.9 to 7.6] | 7.7 [6.6 to 9.1] | 6.4 [5.9 to 7.1] | 6.6 [5.9 to 7.4]
  Day 22: number analyzed (Participants) | 59 | 47 | 49 | 52 | 47 | 40 | 44 | 46
  Day 22 | 49.1 [40.5 to 59.0] | 54.2 [43.8 to 66.8] | 52.7 [43.2 to 65.3] | 56.5 [46.2 to 69.0] | 40.2 [31.4 to 51.5] | 39.7 [28.8 to 49.5] | 44.7 [35.4 to 59.1] | 54.5 [43.3 to 71.5]
  6 months post dose 2: number analyzed (Participants) | 53 | 45 | 44 | 48 | 44 | 36 | 44 | 40
  6 months post dose 2 | 23.7 [19.8 to 27.9] | 26.4 [21.9 to 31.8] | 26.5 [22.2 to 32.4] | 30.8 [25.7 to 36.8] | 25.5 [20.7 to 31.0] | 28.5 [22.3 to 35.0] | 25.3 [20.9 to 31.4] | 29.0 [23.7 to 36.2]

21. Secondary Outcome: GMFR of Serum HI Antibody Titers Against Vaccine-homologous H5N8
Description: as for outcome 2
Time Frame: At Day 22, and 6 months post dose 2 (administered on Day 22)
Population: PPS population. Only those participants with data available at the specified time point have been analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 59 | 47 | 49 | 52 | 47 | 40 | 44 | 46
Ratio
  Day 22 | 9.1 [7.6 to 11.1] | 10.2 [8.3 to 12.6] | 10.2 [8.2 to 12.3] | 10.6 [8.7 to 13.0] | 5.8 [4.5 to 7.5] | 5.1 [4.2 to 7.2] | 6.9 [5.1 to 8.6] | 8.3 [6.3 to 10.4]
  6 months post dose 2: number analyzed (Participants) | 53 | 45 | 44 | 48 | 44 | 36 | 44 | 40
  6 months post dose 2 | 4.3 [3.7 to 5.2] | 5.0 [4.1 to 6.0] | 5.1 [4.2 to 6.1] | 5.8 [4.8 to 6.9] | 3.6 [3.0 to 4.5] | 3.9 [3.2 to 5.0] | 3.8 [3.0 to 4.5] | 4.3 [3.4 to 5.2]

22. Secondary Outcome: Number of Seroprotected Participants for HI Antibody Titers
Description: Seroprotection rate is defined as the number of participants with HI titer value >= 1:40 which is considered as indicating protection.
Time Frame: At Day 1, Day 22, and 6 months post dose 2 (administered on Day 22)
Population: PPS population. Only those participants with data available at the specified timepoint have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 64 | 62 | 59 | 56 | 62 | 56 | 60 | 60
Participants
  Day 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Day 22: number analyzed (Participants) | 59 | 47 | 49 | 52 | 47 | 40 | 44 | 46
  Day 22 | 40 | 40 | 39 | 43 | 25 | 24 | 29 | 33
  6 months post dose 2: number analyzed (Participants) | 53 | 45 | 44 | 48 | 44 | 36 | 44 | 40
  6 months post dose 2 | 14 | 20 | 17 | 25 | 14 | 17 | 13 | 20

23. Secondary Outcome: Number of Seroconverted Participants for HI Antibody Titers
Description: HI seroconversion is defined as a post-vaccination titer >=1:40 in the serum of participants with pre-vaccination titer below 1:10 or as a >=4-fold rise in post-vaccination HI titer with pre-vaccination titer >=1:10.
Time Frame: At Day 22, Day 43 and 6 months post dose 2 (administered on Day 22)
Population: PPS population. Only those participants with data available at the specified timepoint have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 59 | 47 | 49 | 52 | 47 | 40 | 44 | 46
Participants
  Day 22 | 40 | 39 | 39 | 42 | 21 | 21 | 29 | 31
  Day 43: number analyzed (Participants) | 56 | 46 | 47 | 49 | 47 | 40 | 43 | 44
  Day 43 | 55 | 45 | 46 | 49 | 39 | 36 | 40 | 40
  6 months post dose 2: number analyzed (Participants) | 53 | 45 | 44 | 48 | 44 | 36 | 44 | 40
  6 months post dose 2 | 13 | 20 | 17 | 24 | 12 | 14 | 12 | 20

24. Secondary Outcome: Microneutralization (MN) Antibody Titers for a Subset of Participants
Description: Microneutralization testing was performed on 50% of the participants, randomly selected and equally distributed across the different age groups.
Time Frame: At Day 1, Day 22, and 6 months post dose 2 (administered on Day 22)
Population: PPS population subset for MN testing. Only those participants with data available at the specified time points have been analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 32 | 31 | 31 | 26 | 32 | 29 | 29 | 29
Titer
  Day 1 | 5.0 [NA to NA] — 95% CI not calculated as there was no variation in the micro neutralizing titer at visit 1 and it was below level of detection (i.e., below lower limit of quantification) for all participants in this group. | 5.0 [NA to NA] — 95% CI not calculated as there was no variation in the micro neutralizing titer at visit 1 and it was below level of detection (i.e., below lower limit of quantification) for all participants in this group. | 5.0 [NA to NA] — 95% CI not calculated as there was no variation in the micro neutralizing titer at visit 1 and it was below level of detection (i.e., below lower limit of quantification) for all participants in this group. | 5.1 [4.9 to 5.4] | 5.0 [NA to NA] — 95% CI not calculated as there was no variation in the micro neutralizing titer at visit 1 and it was below level of detection (i.e., below lower limit of quantification) for all participants in this group. | 5.2 [4.8 to 5.6] | 5.1 [4.9 to 5.4] | 5.0 [NA to NA] — 95% CI not calculated as there was no variation in the micro neutralizing titer at visit 1 and it was below level of detection (i.e., below lower limit of quantification) for all participants in this group.
  Day 22: number analyzed (Participants) | 30 | 22 | 28 | 25 | 24 | 17 | 21 | 23
  Day 22 | 7.0 [5.6 to 8.6] | 7.8 [6.0 to 10.0] | 8.1 [6.4 to 10.1] | 8.7 [7.0 to 11.3] | 6.4 [5.3 to 7.7] | 5.8 [4.6 to 7.2] | 6.7 [5.5 to 8.3] | 7.0 [5.7 to 8.5]
  6 months post dose 2: number analyzed (Participants) | 26 | 20 | 25 | 24 | 21 | 13 | 21 | 18
  6 months post dose 2 | 6.4 [5.3 to 7.6] | 6.9 [5.6 to 8.5] | 7.0 [5.8 to 8.4] | 6.9 [5.7 to 8.4] | 6.5 [5.3 to 8.0] | 6.2 [4.7 to 8.1] | 6.1 [4.9 to 7.5] | 9.1 [7.2 to 11.4]

25. Secondary Outcome: Number of Seropositive Participants for MN Antibody Titers for a Subset of Participants
Description: A seropositive participant is a participant whose antibody titer is greater than or equal to the assay cut-off value of 1:40.
Time Frame: At Day 1, Day 22, and 6 months post dose 2 (administered on Day 22)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 32 | 31 | 31 | 26 | 32 | 29 | 29 | 29
Participants
  Day 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
  Day 22: number analyzed (Participants) | 30 | 22 | 28 | 25 | 24 | 17 | 21 | 23
  Day 22 | 10 | 10 | 13 | 14 | 5 | 3 | 8 | 8
  6 months post dose 2: number analyzed (Participants) | 26 | 20 | 25 | 24 | 21 | 13 | 21 | 18
  6 months post dose 2 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 10

26. Secondary Outcome: Number of Participants Meeting Vaccine Response (VR) Criteria of MN Antibody Titers for a Subset of Participants
Description: MN VR is defined as titer >=4x LLOQ for participants with pre-vaccination titer below LLOQ or a >=4 -fold increase from pre-vaccination titer for participants with pre-vaccination titer >=LLOQ.
Time Frame: At Day 22, Day 43, and 6 months post dose 2 (administered on Day 22)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 30 | 22 | 28 | 25 | 24 | 17 | 21 | 23
Participants
  Day 22 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1
  Day 43: number analyzed (Participants) | 29 | 21 | 27 | 25 | 24 | 17 | 21 | 21
  Day 43 | 10 | 12 | 10 | 13 | 2 | 6 | 2 | 9
  6 months post dose 2: number analyzed (Participants) | 26 | 20 | 25 | 24 | 21 | 13 | 21 | 18
  6 months post dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

27. Primary Outcome: Number of Participants Reporting pIMDs up to 6 Months Post Dose 2 (Administered on Day 22)
Time Frame: Day 1 to 6 months post dose 2 (administered on Day 22)
Population: The analysis was performed on the Total ES which included participants who received a study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
Number analyzed (Participants) | 66 | 65 | 64 | 63 | 66 | 64 | 66 | 64
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs, MAEs and pIMDs were reported from Day 1 to 6 months post-dose 2 (dose 2 administered on Day 22). Solicited AEs were reported from Day 1 to Day 7 and Day 22 to Day 28 (7 days after each dose). Unsolicited AEs were reported from Day 1 to Day 43.
Arm/Group | Age Group 18-64: FLU Q-PAN H5N8 375_B | Age Group 18-64: FLU Q-PAN H5N8 375_A | Age Group 18-64: FLU Q-PAN H5N8 750_B | Age Group 18-64: FLU Q-PAN H5N8 750_A | Age Group >=65: FLU Q-PAN H5N8 375_B | Age Group >=65: FLU Q-PAN H5N8 375_A | Age Group >=65: FLU Q-PAN H5N8 750_B | Age Group >=65: FLU Q-PAN H5N8 750_A
All-Cause Mortality (participants affected / at risk) | 0/66 | 1/65 | 0/64 | 0/63 | 0/66 | 0/64 | 0/66 | 1/64
Serious Adverse Events (participants affected / at risk) | 1/66 | 1/65 | 0/64 | 2/63 | 2/66 | 2/64 | 2/66 | 2/64
Other Adverse Events (participants affected / at risk) | 50/66 | 40/65 | 40/64 | 50/63 | 39/66 | 44/64 | 34/66 | 41/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Group 18-64: FLU Q-PAN H5N8 375_B (N=66) | Age Group 18-64: FLU Q-PAN H5N8 375_A (N=65) | Age Group 18-64: FLU Q-PAN H5N8 750_B (N=64) | Age Group 18-64: FLU Q-PAN H5N8 750_A (N=63) | Age Group >=65: FLU Q-PAN H5N8 375_B (N=66) | Age Group >=65: FLU Q-PAN H5N8 375_A (N=64) | Age Group >=65: FLU Q-PAN H5N8 750_B (N=66) | Age Group >=65: FLU Q-PAN H5N8 750_A (N=64)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Group 18-64: FLU Q-PAN H5N8 375_B (N=66) | Age Group 18-64: FLU Q-PAN H5N8 375_A (N=65) | Age Group 18-64: FLU Q-PAN H5N8 750_B (N=64) | Age Group 18-64: FLU Q-PAN H5N8 750_A (N=63) | Age Group >=65: FLU Q-PAN H5N8 375_B (N=66) | Age Group >=65: FLU Q-PAN H5N8 375_A (N=64) | Age Group >=65: FLU Q-PAN H5N8 750_B (N=66) | Age Group >=65: FLU Q-PAN H5N8 750_A (N=64)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 4 (5) | 4 (4) | 6 (11) | 7 (8) | 4 (4) | 5 (7) | 4 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 11 (13) | 8 (8) | 8 (9) | 6 (8) | 3 (3) | 2 (2) | 5 (6) | 4 (4)
Nausea (Gastrointestinal disorders) | 12 (13) | 8 (8) | 4 (4) | 9 (15) | 5 (6) | 4 (5) | 5 (6) | 4 (6)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 7 (9) | 9 (9) | 4 (4) | 8 (8) | 5 (6) | 3 (3) | 1 (1) | 4 (5)
Fatigue (General disorders) | 29 (43) | 21 (28) | 19 (25) | 24 (31) | 11 (14) | 16 (25) | 9 (10) | 15 (20)
Fever (General disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 4 (4) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 5 (7)
Injection site pain (General disorders) | 44 (70) | 37 (53) | 33 (48) | 41 (62) | 27 (40) | 25 (36) | 18 (26) | 31 (44)
Injection site swelling (General disorders) | 5 (5) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 1 (2) | 0 (0) | 5 (7)
Sweating (General disorders) | 12 (15) | 8 (10) | 5 (6) | 10 (12) | 7 (10) | 3 (4) | 2 (2) | 4 (5)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (20) | 14 (16) | 5 (6) | 11 (15) | 5 (5) | 9 (10) | 6 (7) | 8 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 29 (40) | 25 (33) | 17 (25) | 30 (41) | 12 (15) | 15 (19) | 8 (11) | 17 (23)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain fog (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 30 (39) | 15 (18) | 12 (14) | 18 (25) | 10 (14) | 13 (16) | 8 (10) | 13 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT05975840/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT05975840/SAP_001.pdf